CLINICAL TRIAL: NCT02718287
Title: Evaluation of the Home Visiting Pilot Programa Cresça Com Seu Filho (PCCSF) on Early Childhood Outcomes: a Cluster-Randomized Trial in Fortaleza Brazil
Brief Title: Evaluation of the Home Visiting Pilot Program on Early Childhood Outcomes in Fortaleza Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inter-American Development Bank (Other)
Collaborators: Municipal Secretary of Health, Fortaleza Brasil (Unknown); Universidade Federal do Ceara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IDB-2016-BR-1
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Child Development
Keywords: language development; socio-emotional development; cognitive development; motor skills
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment: (Experimental): Home visiting with PCCSF
  Interventions: Behavioral: Home visiting intervention PCCSF (220 clusters)
- Control (Experimental): Home visiting no PCCSF
  Interventions: Behavioral: Home visiting without PCCSF (220 clusters)

INTERVENTIONS:
Behavioral: Home visiting intervention PCCSF (220 clusters) — Low income mothers of children 0-2.5 years of age in the randomized treatment micro-areas will receive home visits by community health workers trained in the PCCSF curriculum in addition to the basic health curriculum. The community health workers are supervised by trained and experienced nurses.
  Arms: Treatment:
Behavioral: Home visiting without PCCSF (220 clusters) — Low income mothers of children 0-2.5 years of age in the randomized control micro-areas will receive home visits by community health workers trained in the standard basic health curriculum (no PCCSF).
  Arms: Control

SUMMARY:
This is a cluster-randomized study of a home visiting program targeting mothers of children 0 to 2.5 years of age with the objective of improving global child development. The program, Programa Cresça com Seu Filho (PCCSF), will be randomized across 220 microareas in the poorest Region (V) of the state of Fortaleza, Brazil.

DETAILED DESCRIPTION:
This is an evaluation of pilot program, Programa Cresça com Seu Filho (PCCSF) which is publically funded and, developed in a partnership between the Ministry of Health (MoH) of Brazil and the municipal government of Fortaleza. The program targets low-income mothers of children 0 to 2.5 years old, living in low-income neighborhoods in Fortaleza Brazil. The home visits are carried out by community health workers (CHW), who currently work for the Ministry of Health as part of the program Programa Saúde da Família. The CHWs will be trained on the PCCSF curriculum in order to provide 1-hour visits with the early stimulation package during two years. The PCCSF home visiting program is planned to begin implementation the week of March 15, 2016 for half of the community health workers and April 15, 2016 for the other half.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children ages 0-2.5 years of age
* Included in the poverty registry CadastroUnico
* Residents of specific 440 poor microareas of Region V of Fortaleza

Exclusion Criteria:

* Data will not be collected if parental consent not given.

Ages: 1 Day to 28 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2520 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Denver Developmental Screening Test II- aggregate rating of language skills | change from baseline to follow-up at 18 months
  language development
Denver Developmental Screening Test II - aggregate rating of socioemotional skills | change from baseline to follow-up at 18 months
  socioemotional development
Denver Developmental Screening Test II -aggregate rating motor skills | change from baseline to follow-up at 18 months
  motor development
Denver Developmental Screening Test II -aggregate rating cognitive skills | change from baseline to follow-up at 18 months
  cognitive development

CONTACTS AND LOCATIONS:
Overall Officials: Florencia Lopez Boo, Ph.D., Principal Investigator — Inter-American Development Bank; Cristiana Ferreira da Silva, Ph.D., Principal Investigator — Secretaria Municipal de Saúde de Fortaleza; Marcia Rocha, M.A., Principal Investigator — Inter-American Development Bank; Suzanne Duryea, P.h.D., Principal Investigator — Inter-American Development Bank